CLINICAL TRIAL: NCT04906811
Title: Prospective Comparison of the Revolve™ and AuraGen 1-2-3™ With AuraClens™ Systems in Processing of Lipoaspirate for Autologous Fat Grafting to the Breast
Brief Title: Prospective Comparison of Revolve™ and AuraGen 123 With AuraClens™ in Autologous Fat Grafting to the Breast
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study discontinued due to lack of subject follow-up.
Sponsor: AuraGen Aesthetics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AUGCS001
Record Dates: First submitted 2021-05-20; First posted 2021-05-28 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Autologous Fat Grafting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Fat grafting with the AuraGen 1-2-3 with AuraClens System (Active Comparator): Patients undergoing an aesthetic fat grafting procedure to the breast without a breast implant. Lipoaspirate processed with the AuraGen 1-2-3 with AuraClens system.
  Interventions: Device: AuraGen 1-2-3 with AuraClens system (BK190433)
- Fat grafting with the Revolve System (Active Comparator): Patients undergoing an aesthetic fat grafting procedure to the breast without a breast implant. Lipoaspirate processed with the Revolve System.
  Interventions: Device: Revolve System (K120902)

INTERVENTIONS:
Device: AuraGen 1-2-3 with AuraClens system (BK190433) — Fat grafting to the breast in patients undergoing an aesthetic procedure without a breast implant. Device used: AuraGen 1-2-3 with AuraClens system
  Arms: Fat grafting with the AuraGen 1-2-3 with AuraClens System
Device: Revolve System (K120902) — Fat grafting to the breast in patients undergoing an aesthetic procedure without a breast implant. Device used: Revolve System
  Arms: Fat grafting with the Revolve System

SUMMARY:
The purpose of this study is to compare fat graft retention over time from lipoaspirate processed using two FDA-cleared devices: the Revolve System (K120902) and the AuraGen 1-2-3 with AuraClens Lipoaspirate Wash System (BK190433).

DETAILED DESCRIPTION:
This is a single-center, prospective, randomized study enrolling patients undergoing an aesthetic fat grafting procedure to the breast without a breast implant. A total of 20 patients will be enrolled in the study. Ten patients will receive lipoaspirate processed with the Revolve and ten patients will have lipoaspirate processed with the AuraGen 1-2-3 with AuraClens.

Patients will be followed on post-procedure months 3, 6, and 12. Fat graft retention will be evaluated by photographic assessment by blinded reviewers, and 3D imaging. Patient satisfaction will be measured using the Breast-Q - Augmentation survey.

ELIGIBILITY:
Inclusion Criteria:

* Female patients > 18 years and < 65 years of age
* Patients undergoing an aesthetic fat grafting procedure to the breast (breast augmentation) without a breast implant.
* Patients must be able to provide written informed consent, understand and be willing to comply with study-related procedures and follow-up visits.
* Patients must be non-smokers.
* Patients with available/adequate harvest sites for fat grafting.
* Anticipated harvested fat volume between 400 and 1400 cc
* Anticipated fat injection volume 150-350 cc per breast
* Patients must agree to maintain their weight (i.e. within 5%) by not making any major changes in their diet or lifestyle during the study.

Exclusion Criteria:

* Skin rash in the treatment area.
* Patients who smoke or use nicotine products.
* Patients with bleeding disorders or currently taking anticoagulants.
* Patients with a history of trauma or surgery to the treatment area.
* Patients with a history of breast cancer.
* Active, chronic, or recurrent infection.
* Compromised immune system (e.g. diabetes).
* Hypersensitivity to analgesic agents.
* Co-morbid conditions that could limit their ability to participate in the study or to comply with follow-up requirements.
* Untreated drug and/or alcohol abuse.
* Pregnant or breastfeeding.
* Any issue that, at the discretion of the investigator, would contraindicate the patient's participation.
* Patients who do not wish to have the study area (breast) photographed

NOTE Please note that there is no remuneration for participation in this study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients
Enrollment: 17 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2024-02-12 (Actual); Study Completion 2024-02-12 (Actual)

PRIMARY OUTCOMES:
Fat volume retention at 3 months post-op | 3 months post-op
  Measurement of volume of fat graft at 3 months post-op, using 3D photography
Fat volume retention at 6 months post-op | 6 months post-op
  Measurement of volume of fat graft at 6 months post-op, using 3D photography
Fat volume retention at 12 months post-op | 12 months post-op
  Measurement of volume of fat graft at 6 months post-op, using 3D photography

SECONDARY OUTCOMES:
Patient Satisfaction | 3 months post-op
  Breast-Q - Augmentation Survey
Patient Satisfaction | 6 months post-op
  Breast-Q - Augmentation Survey
Patient Satisfaction | 12 months post-op
  Breast-Q - Augmentation Survey

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A Del Vecchio, MD, Principal Investigator — Back Bay Plastic Surgery
Locations (1):
- Back Bay Plastic Surgery, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Both devices are FDA-cleared. This is a marketing study.